CLINICAL TRIAL: NCT06116500
Title: A Modified Removable Orthodontic Appliance for Maxillary Expansion and Treatment of Class II Malocclusion: A Randomized Clinical Trial
Brief Title: Effectiveness of Modified Functional Appliance With Expander
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of Baghdad (Other)
Responsible Party: Principal Investigator, Anosh Aram Haik, Principal investigator, University of Baghdad
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 664422
Record Dates: First submitted 2023-10-21; First posted 2023-11-03 (Actual); Last update posted 2023-11-07 (Actual); Status verified 2023-10

CONDITIONS: Class II Malocclusion
Keywords: twin block; thermoplastic material; clear expander,; adolescent; clinical trial
MeSH Terms: conditions — Overbite

STUDY DESIGN:
Intervention Model Description: The patients will be treated with twin block appliance
Who Masked: Participant
Masking Description: In the study, data collection and measurement will be conducted with the investigator. However, it won't be possible to blind the operator (investigator) due to the appliance design/shape difference, making the study single-blinded. Each patient will not know which type of twin block appliance will be used for them.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Modified twin block appliance with expander group (Experimental): For 24 patients with class II division malocclusion in their growing stages, using a 2 mm biocompatible and rigid PET-G thermoforming material to create two clear appliances for each patient. The material will be adapted separately on maxillary and mandibular casts using a pressure molding vacuum machine. Then, the appliances will be trimmed and finished and transferred to the articulator with the aid of a pre-existing working wax bite. The ramps will be made of cold cure acrylic on the thermoplastic sheets. Next, the expansion screw will be placed in the midline of the maxillary cast, and the maxillary appliance will be split midpalatally to fit the patient's individual needs.
  Interventions: Device: Modified twin block appliance with expander; Device: Conventional twin block appliance with expander
- Conventional twin block appliance with expander group (Experimental): For 24 patients in a growing stage with class II division 1 malocclusion, these appliances will consist of removable maxillary and mandibular appliances. These will have a labial bow, Adam's clasps on the first molars, ball end clasps with incisal capping and expansion screw. The inclined bite blocks (ramps) will act as a guide to move the mandible forward.
  Interventions: Device: Modified twin block appliance with expander; Device: Conventional twin block appliance with expander

INTERVENTIONS:
Device: Modified twin block appliance with expander — These appliances are myofunctional appliance used for treating class II division growing adolescents.
Device: Conventional twin block appliance with expander — These appliances are myofunctional appliances used for treating class II division growing adolescents.

SUMMARY:
This clinical trial compares the effectiveness of a myofunctional appliance that uses a clear and modified twin block appliance with an expander made from 2mm biocompatible polyethylene terephthalate modified with Glycol thermoplastic material with a conventional twin block appliance with an expander. The trial will be conducted on adolescent patients with class II division 1.

DETAILED DESCRIPTION:
In a multicenter single-blinded randomized clinical trial study with two-arm parallel groups, a computer random generator will develop a simple randomization with an equal allocation ratio (1:1) and without stratification. The investigator will initially assess the patients for eligibility to be included in the study. Those who will meet the inclusion criteria, the parents will be informed about the nature of the study verbally to get the initial approval for participation. Then they will be provided with the patient information sheet and consent form.

According to the sample size calculation, 48 patients will be recruited (24 for each group), and impressions and lateral cephalometric radiography will be taken before treatment and bite registration then the appliance inserted, and the patient will be checked every two weeks for expansion and every four weeks for overjet recording. The treatment will be continuing for 6 months to take final records. The collected data will include cephalometric evaluation, clinical evaluation, scanned upper model evaluation, and finally patient satisfaction from the appliance.

Data will be analyzed using Statistical Package for Social Sciences for Windows, version 26.0 including descriptive statistic (number, mean, and standard deviation), Reliability statistic (interclass correlation coefficient), and Inferential statistics (independent samples t-test).

ELIGIBILITY:
Inclusion Criteria:

1. Patients' age at the start of treatment: at growth spurt [in stage 2 (Acceleration) - 3 (Transition) of cervical vertebral maturation].
2. Skeletal and dental relationships: skeletal class II with normal maxilla and retrognathic mandible. Moderate to severe dental class II division 1 malocclusion with overjet ≥ 8 mm.
3. Horizontal/normal growth pattern.
4. Convex profile with decreased or normal lower facial height (clinically and radiographically).
5. Well-aligned/mild crowding of maxillary and mandibular dental arches.
6. Good oral health free from caries and periodontal problems at the start of treatment.

Exclusion Criteria:

1. Patients with vertical growth pattern or backward mandibular rotation tendency.
2. Patients with open bite
3. Patients with obvious facial asymmetry.
4. Patients with orofacial clefting.
5. Patients with bad oral habits.
6. Active periodontal disease.

Ages: 10 Years to 13 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 48 (Estimated)
Dates: Start 2023-05-09 (Actual); Primary Completion 2024-05-09 (Estimated); Study Completion 2024-06-09 (Estimated)

PRIMARY OUTCOMES:
Anteroposterior skeletal changes | T0 (before treatment), T1 (at end of the study) around 6-9 months
  Skeletal changes using cephalometric radiographs including different angular measurements to estimate the changes between dental bases before and after treatment.
Vertical skeletal changes | T0 (before treatment), T1 (at end of the study) around 6-9 months.
  Skeletal changes using cephalometric radiographs including different linear measurements to estimate the changes between dental bases before and after treatment.

SECONDARY OUTCOMES:
Soft tissue change | T0 (before treatment), T1 (at end of the study) around 6-9 months
  Measurements using cephalometric radiographs including different angular measurements to estimate the soft tissue changes before and after treatment.
Dentoalveolar changes | T0 (before treatment), T1 (at end of the study) around 6-9 months
  Measurements using cephalometric radiographs include different angular measurements to estimate the changes between teeth before and after treatment.
Study model evaluation | T0 (before treatment), T1 (at end of the study) around 6-9 months.
  The scanned upper study model will be used to calculate the amount of expansion before and at the end of the study.
Patient satisfaction from the appliance | around 4 months.
  Patient satisfaction with both appliances will be estimated using a questionnaire at the middle of treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Yassir A Yassir, Ph.D. (UK), Study Chair — Baghdad University, Collage of Dentistry
Locations (1):
- University of Baghdad, Collage of Dentistry, Baghdad, Al-Rusafa, Bab Al-moadham, Iraq

REFERENCES:
- [Derived] Haik AA, Yassir YA. Efficiency of Polyethylene Terephthalate Glycol Thermoplastic Material to Functional and Expansion Forces in Orthodontic Applications: An Experimental Study. ScientificWorldJournal. 2025 Jan 10;2025:7232779. doi: 10.1155/tswj/7232779. eCollection 2025. PMID 39840371